CLINICAL TRIAL: NCT06858215
Title: African Youth in Mind (Y-MIND) - Pilot Feasibility Trial of a Brief Psychological Intervention for Young People Aged 15-24 with Depression in Zimbabwe
Brief Title: African Youth in Mind (Y-MIND) - Pilot Feasibility Trial of a Brief Psychological Intervention for Young People with Depression in Zimbabwe
Acronym: Y-MIND
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University of Zimbabwe (Other); University of Ghana (Other); Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR/DP-23/24-44227; NIHR133384 (Other Grant/Funding Number: National Institute for Health and Care Research)
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Depression
Keywords: depression; psychological therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Y-MIND Intervention (Experimental): All participants in the intervention arm will receive the the Y-Mind intervention. Y-Mind intervention will be delivered by trained and supervised lay counsellors in primary health care clinics. The six sessions will include a) psychoeducation on depression, b) behavioural activation (helping the participant see the connection between their behaviour, daily activities, and low mood and activity scheduling) and c) problem-solving therapy (the counsellor helps the participant identify and define a specific problem to work on, evaluate the potential solutions to the problem, and carry out the selected solution(s)).
  Interventions: Behavioral: Y-MIND Intervention

INTERVENTIONS:
Behavioral: Y-MIND Intervention — All participants in the intervention arm will receive the the Y-Mind intervention. Y-Mind intervention will be delivered by trained and supervised lay counsellors in primary health care clinics. The six sessions will include a) psychoeducation on depression, b) behavioural activation (helping the participant see the connection between their behaviour, daily activities, and low mood and activity scheduling) and c) problem-solving therapy (the counsellor helps the participant identify and define a specific problem to work on, evaluate the potential solutions to the problem, and carry out the selected solution(s)).

SUMMARY:
The overarching aim of this single-arm pilot study is to assess the feasibility of implementing a psychological intervention (Y-MIND), delivered by lay counsellors, for the treatment of depression among young people aged 15-24 in in Harare Province, Zimbabwe. The study aims to assess the feasibility, acceptability and fidelity of delivering the six-session Y-MIND intervention, and collect preliminary clinical outcomes for depression at 5-month follow up.

DETAILED DESCRIPTION:
The overarching aim of this single-arm pilot study is to assess the feasibility of implementing a psychological intervention (Y-MIND) for the treatment of depression among young people aged 15-24 in in Harare Province, Zimbabwe. The six session problem solving therapy intervention will be delivered by trained and supervised lay counsellors. 50 young people will be recruited aged 15-24 through primary care clinics to receive the Y Mind intervention. The study aims to assess the feasibility, acceptability and fidelity of delivering the six-session Y-MIND intervention, and collect preliminary clinical outcomes for depression at 5-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Young people aged 15-24 years
* Scoring 11 or more on the locally validated Patient Health Questionnaire-9 (PHQ-9) for those aged 18+ and 10 or more on the Patient Health Questionnaire Adolescent (PHQ-A) for those < 18 years.
* Willing and able to be followed up for 5 months.
* Willing and able to provide informed consent if aged 18+, or, if aged below 18, willing and able to give informed assent and to approach a caregiver for informed consent procedures

Exclusion Criteria:

* Currently receiving any psychological treatment for any common mental disorder through formal health care services
* Active major mental disorder, advanced physical illness which would interfere with their ability to take part in the study or are actively suicidal (assessed through screening using the P4 screener).
* Those with visual and/or hearing impairment; defined as being unable to see and read the intervention manual or hear the interventionist sitting approximately 1 metre away. This will be assessed at informed consent procedures.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2025-08-02 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention | At the end of treatment (week 6) (or at their 5 months post baseline assessment if the treatment sessions were not attended)
  Feasibility of the intervention, defined as extent to which the Y Mind intervention can be successfully delivered by interventionists to reduce symptoms of depression in young people, will be measured using the 'Feasibility of Intervention Measure' (FIM) with adolescents who received the Y-MIND intervention.

SECONDARY OUTCOMES:
Symptoms of depression | 5 months post baseline assessment
  Symptoms of depression at 5 months post baseline assessment measured using the PHQ-9. The mean PHQ-9 score will be summarised at baseline and 5 month follow up. This will allow for calculation of sample size for a future definitive trial.
Acceptability of the intervention | At end of Y-MIND intervention sessions or at 5 months post baseline assessment
  Acceptability, defined as the extent to which the programme is perceived to be agreeable and acceptable to treat depression and adolescents, will be measured using the Acceptability of Intervention Measure (AIM) with adolescents at the end of their last intervention session, (or at their 5 month follow up if the intervention session was not attended), and with lay counsellors when they finish delivering the intervention. It will also be explored through semi-structured interviews with young people (at end of 5 months post baseline assessment) and focus group discussions with lay counsellors (after they have finished delivering all intervention sessions).
Feasibility of the intervention (lay counsellors) | At the end of treatment (week 6) (or at their 5 months post baseline assessment if the treatment sessions were not attended)
  Feasibility of the intervention, defined as extent to which the Y Mind intervention can be successfully delivered by interventionists to reduce symptoms of depression in young people will be measured using the Feasibility of Intervention Measure (FIM) (Weiner et al. 2017) with lay counsellors when they finish delivering the intervention and using semi-structured interviews with adolescents and focus group discussions with lay counsellors
Fidelity to delivering the psychological intervention | From the first treatment session (week 1) to the end of treatment (week 6)
  Fidelity to delivering the psychological intervention, defined as the extent to which the intervention was delivered as intended, and measured by rating 20% of audio-recorded psychological intervention sessions using a culturally adapted form of ENACT called the 'Problem-Solving Therapy Fidelity Scale (PROOF)' tool. Fidelity of receipt of the psychological intervention, defined as the extent to which the intervention is received as intended and measured by recording session attendance.
Symptoms of anxiety | 5 months post baseline assessment
  Symptoms of anxiety at 5 months post baseline assessment measured using the GAD-7. The mean GAD-7 score will be summarised at baseline and 5 month follow up. This will allow for calculation of sample size for a future definitive trial.
Appropriateness of the intervention | At end of Y-MIND intervention sessions or at 5 months post baseline assessment
  Appropriateness, defined as the extent to which the programme is perceived as being relevant to treat depression in adolescents, will be measured by using the Intervention Appropriateness Measure (IAM) with adolescents at the end of their last intervention session, (or at their 5 month follow up if the intervention session was not attended) and with guidance and counselling coordinators when they finish delivering the intervention. It will also be explored through semi-structured interviews with young people (at end of 5 months post baseline assessment) and focus group discussions with lay counsellors (after they have finished delivering all intervention sessions).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zimbabwe, Harare, Zimbabwe